CLINICAL TRIAL: NCT02356614
Title: A Post-approval LAP-BAND® Lower Body Mass Index (LBMI) Study
Status: Terminated | Type: Observational
Why Stopped: Terminated is based on the availability of long-term safety and effectiveness data from the OSB Lead-HERo-002 study and published literature.
Sponsor: Apollo Endosurgery, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Apollo-001
Record Dates: First submitted 2015-02-02; First posted 2015-02-05 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-03

CONDITIONS: Obesity; Overweight
Keywords: Lap Band
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a post-approval, multicenter, prospective, non-randomized, open-label, clinical study to evaluate the safety and effectiveness of the LAP-BAND® AP System in a lower obese population (BMI ≥ 30 kg/m2 and < 40 kg/m2) with one or more obesity-related comorbidity up to 10 years after implantation.

The reason your study has been terminated is based on the availability of long-term safety and effectiveness data from the OSB Lead-HERo-002 study and published literature.

DETAILED DESCRIPTION:
FDA post-approval study designed to collect prospective data in a real-world setting to evaluate long-term safety and effectiveness of the LAP BAND® System in patients with a BMI of ≥ 30 kg/m2 and < 40 kg/m2 and one or more comorbid conditions. The Apollo-001 Study is a prospective, 10 year, multicenter study of patients who have decide to undergo implantation of the LAP-BAND AP® system. Outcomes include device explants, changes in weight, comorbid condition status, device- and procedure-related AEs, and reoperations.

The LBMI study was part of the condition of approval (CoA) for the Lap-Band device. It was terminated because it was no longer required to fulfill the condition of approval for the device. Apollo was able to fulfill the condition of approval (CoA) for the Lap-Band device by using data from published literature and another recently completed study (OSB Lead-Hero-002 study) which had long-term safety and effectiveness data addressing the conditions of approval.

ELIGIBILITY:
Inclusion Criteria:

1. LAP-BAND® System placed in a facility in the United States
2. BMI ≥ 30 kg/m2 and < 40 kg/m2 prior to LAP-BAND® placement
3. Presence of 1 or more obesity-related comorbidities prior to LAP-BAND® placement
4. Aged 18 or older

Exclusion Criteria:

1. Prior bariatric surgery.
2. Participating in another ongoing clinical study in which concomitant diagnostic or therapeutic intervention that would reasonably be expected to alter patterns of care, use of medications or the outcomes under study.
3. Vulnerable patients or those unable to exercise free informed consent.
4. Inability to complete the questionnaires.
5. Patients who are addicted to alcohol and/or drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese adult patients with a BMI ≥ 30 kg/m2 and < 40 kg/m2 with one or more comorbid conditions that have had a LAP-BAND® System implanted.
Sampling Method: Non-Probability Sample
Enrollment: 325 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-03-08 (Actual); Study Completion 2018-03-08 (Actual)

PRIMARY OUTCOMES:
Percentage of Explants | 5 Years
  The primary objective is to assess the percentage of patients who experience an explant of the LAP BAND System within 5 years of implantation.

SECONDARY OUTCOMES:
Response to the LAP-BAND | 5 Years
  Secondary objectives include assessment of patients who respond to the LAP BAND® System at 5 years, where response is defined as achieving at least 7%Total Body Loss (TBL), assessment of prevalence of diabetes at 5 years, and assessment of changes in obesity-related comorbid conditions at 5 years.
Diabetes | 5 Year
  Assessment of prevalence of diabetes at 5 years
Obesity related Comorbidity | 5 Year
  Assessment of changes in obesity-related comorbid conditions at Year 5

OTHER OUTCOMES:
Percent Reoperations, Esophageal Dilatation, esophageal dysmotility, and related adverse events | 10 Years
  Percentage of patients experiencing reoperations, esophageal dilatation, esophageal dysmotility, and other device-related and procedure-related adverse events observed over the study assessment period.

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Naveira, Study Director — Apollo Endosurgery, Inc.
Locations (11):
- United States (11):
  - Surgical Associates, Fountain Valley, California
  - Illinois Bariatric Center, Champaign, Illinois
  - Bariatric Institute of Greater Chicago, Chicago, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - Louisville Surgical Associates, Louisville, Kentucky
  - Surgical Specialists of Louisiana, Metairie, Louisiana
  - Advanced Weight Loss Surgery, Rockville, Maryland
  - St. Alexius New Start, St Louis, Missouri
  - New York University, New York, New York
  - Center for Metabolic & Bariatric Surgery, Cincinnati, Ohio
  - Utah Lap Band and General Surgery, Draper, Utah